CLINICAL TRIAL: NCT00222131
Title: Inhibition of Gastric Acid Is the Key To Satisfactory Relief of Symptoms and Restoration of the Quality of Life in Patients With Epigastric Pain Related to Non-Ulcer Dyspepsia During Therapy With Esomeprazole
Brief Title: Inhibition of Gastric Acid is the Key to Satisfactory Relief of Symptoms With Esomeprazole in NUD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 8777
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Indigestion
Keywords: Epigastric Pain; Non-Ulcer Dyspepsia (NUD)
MeSH Terms: conditions — Dyspepsia | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- 2 (Active Comparator): Esomeprazole
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — Esomeprazole 40 mg QD
  Other Names: Nexium
  Arms: 2
Other: Placebo — Placebo
  Arms: 1

SUMMARY:
Inhibition of gastric acid is the key to satisfactory relief of symptoms with esomeprazole in NUD patients

DETAILED DESCRIPTION:
Enrolled patients will undergo 24h gastric pH monitoring and subsequently (if gastric pH drops below pH 4 during 24h monitoring) will be randomized to receive placebo (40 mg QD) or esomeprazole (40 mg QD) for 16 weeks of therapy. 24h gastric pH monitoring will be repeated 2nd and 3rd time in all participating patients at the end of 4th and 8th weeks of therapy. Additionally, in all participants NUD symptoms will be re-assessed at the end of 4th, 8th, 12th and 16th weeks of therapy.

ELIGIBILITY:
Inclusion criteria:

A. Males and females of age 18-55. B. A diagnosis of epigastric pain/discomfort (located in the upper abdomen) rated by the patient as moderate to severe in intensity (on a four-point categorical scale), which has been present at least 3 times per week for 12 weeks, unrelated to exercise.

C. Patients may have other symptoms of NUD including heartburn, regurgitation, bloating (abdominal distension), early satiety (feeling of fullness), belching (burping), or nausea; however, the dominant symptom must be epigastric pain/discomfort.

D. Capable of and willing to give informed consent and comply with all study requirements.

Exclusion criteria:

A. H. pylori positive serology. B. Regular use of NSAIDs or more than 100 mg of aspirin. C. Patients requiring chronic treatment with any medication inducing GI symptoms (e.g., certain antibiotics, codeine, etc.).

D. History or presence of endoscopic/radiological evidence of esophagitis. E. History or presence of chronic gastric or duodenal ulcer. F. History or presence of duodenal erosions. G. History or previous upper GI surgery. H. Presence of concomitant symptoms of irritable bowel syndrome (IBS) as assessed by three or more of the Manning or Rome criteria.

I. History or presence of other known organic disease that might explain the dyspepsia symptoms (e.g., symptomatic gallstones).

J. Pregnancy or lactation. K. Inadequate contraception. L. Regular consumption of greater than 2 fluid ounces of beverage alcohol (corresponding to 2 cocktails or 40 fluid ounces of beer or 16 fluid ounces of wine) per day.

M. History of substance abuse. N. Unwillingness or expected inability to tolerate absence of antisecretory medications (antacids, H2 receptor antagonists or Proton pump inhibitors (PPIs) or other GI pharmacotherapy for a period of time of study protocol (16 weeks maximum).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2003-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mccallum, MD, Principal Investigator — University of Kansas Medical Center; Jerzy Sarosiek, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Esomeprazole: Esomeprazole 40 mg one time a day (QD)
- Placebo: Matching placebo
Period: Overall Study
Arm/Group | Esomeprazole | Placebo
Started | 38 | 35
Completed | 38 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole | Placebo | Total
Number analyzed (Participants) | 38 | 35 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 35 | 73
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 17 | 15 | 32
Region of Enrollment [Number; unit: participants]
  United States | 38 | 35 | 73

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Satisfactory Relief of Non-ulcer Dyspepsia Symptoms
Description: Dyspeptic symptoms severity will be assessed with validated 7-graded diary cards. The diary cards asked "Please state for each day if you have experienced pain or discomfort in the stomach." Measure taken over 7 consecutive days of a 2 week run in and at the end of each therapeutic period.
Time Frame: 8 Weeks
Measure: Number; unit: percentage of participants
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 38 | 35
percentage of participants
  4 Weeks | 71 | 34
  8 Weeks | 82 | 56

2. Secondary Outcome: Satisfactory Relief of Non-ulcer Dyspepsia Symptoms as Time Gastric pH Remained > 4.0 Within 24 Hours
Description: Time (minutes) gastric pH remained >4.0 during 24-hours gastric pH monitoring.
Time Frame: 8 Weeks
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Esomeprazole | Placebo
Number analyzed (Participants) | 38 | 35
minutes
  4 Weeks | 1170 (51.6) | 905 (134.8)
  8 Weeks | 1050 (74.3) | 762 (101.8)

ADVERSE EVENTS:
Arm/Group | Esomeprazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/35
Other Adverse Events (participants affected / at risk) | 0/38 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes